CLINICAL TRIAL: NCT03384056
Title: Comparison of Air-Q Self Pressurized Airway Device With Blocker With Proseal Laryngeal Mask Airway in Anesthetized Paralyzed Adult Female Patients Undergoing Elective Gynecological Operations
Brief Title: Respiration and The Airway With Supraglottic Airway Devices
Status: Completed | Type: Observational
Sponsor: Reham Ali Abdelhaleem Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Reham Ali Abdelhaleem Abdelrahman, Anaesthesia Lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: AR-1974
Record Dates: First submitted 2017-12-14; First posted 2017-12-27 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Laryngeal Masks Comparison

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Self Pressurized Airway Device with Blocker
  Interventions: Device: Self Pressurized Airway Device with Blocker
- Proseal Laryngeal Mask Airway
  Interventions: Device: Proseal Laryngeal Mask Airway

INTERVENTIONS:
Device: Self Pressurized Airway Device with Blocker — used in adult low risk females undergoing elective gynecological operations
  Groups: Self Pressurized Airway Device with Blocker
Device: Proseal Laryngeal Mask Airway — used in adult low risk females undergoing elective gynecological operations.
  Groups: Proseal Laryngeal Mask Airway

SUMMARY:
The investigators aim to compare the airway seal pressure( oropharyngeal leak pressure) of the Self Pressurized Airway Device with Blocker® with the ProsealTM Laryngeal Mask Airway (P-LMA)in anesthetized paralyzed adult female patients undergoing elective gynecological operations. The investigators aim at assessment of fitting of both devices against the glottic region that detected by the flexible fiberoptic bronchoscope( Pentex Corporation, Medical Division, Singapore)and assessment of any associated postoperative complications.

Hypothesis:

The investigators hypothesize that the self-pressurized air-Q with blocker has a greater seal pressure compared to Proseal, easier and faster in insertion with less morbidity and complications during and after its insertion.

DETAILED DESCRIPTION:
The study will be carried on adult female patients to reduce variability in size of the chosen device to enable the investigators to analyze the performance parameters of the two devices with greater authority. The study will be done on anesthetized paralyzed adult female patients undergoing elective gynecological operations that require neuromuscular block but not necessarily tracheal intubation. The investigators will recruit 150 adult female(18-55 years old, ASAI&II) patients to a prospective randomized comparative controlled two-arm parallel clinical trial. Patients with history of upper respiratory tract infections, obstructive sleep apnea, potentially full stomach (trauma, morbid obesity BMI> 35, pregnancy, history of gastric regurgitation and heart burn), those with esophageal reflux (hiatus hernia), and those of coagulation disorders will be excluded from the study. All patients will be assessed pre-operatively El-Ganzouri airway score to assess the expected difficulty of intubation and patients with airway scores ≥ 5 will be excluded from the study. The patients will be randomly allocated into two groups(the SP-Blocker group & the P-LMA group; each group is 75 patients) using computer generated program . An online randomization program (http://www.randomizer.org) will be used to generate random list and to allocate patients into the study groups. Random allocation numbers will be concealed in opaque closed envelops. The patient and investigator assessing study outcomes will all be blinded to the study groups allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients ASA I&II
* Age: 18- 55 years old
* BMI < 35
* Undergoing elective gynecological operations.

Exclusion Criteria:

* Patients with history of upper respiratory tract infections and obstructive sleep apnea.
* Patients who are potentially full stomach such as trauma, pregnancy, history of gastric regurgitation &heart burn, those with esophageal reflux or hiatus hernia.
* Patients with coagulation disorders.
* Patients with El-Ganzouri airway score ≥ 5 will.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adult female patients undergoing elective gynecological operations.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
airway seal pressure | one year
  pressure at which leak starts to occur
fitting of the device against larynx | one year
  detected by the flexible fiberoptic

SECONDARY OUTCOMES:
insertion time of the device | one year
  is defined as time in seconds from the chosen device touching the teeth to the first recorded near rectangular capnogram curve in the presence of satisfactory bilateral chest expansion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Surgical ICU, and Pain Management, Cairo, Egypt